CLINICAL TRIAL: NCT06805279
Title: Comparing Axillary Vein Cannulation with 'Hockey' Probe Versus Linear Probe for Central Venous Access
Brief Title: Axillary Vein Cannulation: 'Hockey' Probe Versus Linear Probe
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: KB/27/2022
Record Dates: First submitted 2024-12-30; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-12

CONDITIONS: CVC; Ultrasound Guided Central Venous Cannulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Hockey ultrasound probe: Use of Hockey ultrasound probe for axillary vein cannulation
  Interventions: Procedure: Axillary Vein Cannulation
- Linear ultrasound probe: Use of linear ultrasound probe for axillary vein cannulation
  Interventions: Procedure: Axillary Vein Cannulation

INTERVENTIONS:
Procedure: Axillary Vein Cannulation — This study aims to evaluate the potential advantages of using the "hockey stick" ultrasonography probe for axillary vein cannulation and determine whether this probe enhances axillary vein imaging, accelerates the central vein cannulation procedure and reduces the rate of complications compared to the linear probe

SUMMARY:
Central venous catheterization, specifically through the axillary vein, is a procedure of critical importance in various clinical contexts. Site selection is dependent on clinical assessment, experience and the physician preference. This study aims to evaluate the potential advantages of using the "hockey stick" ultrasonography probe for axillary vein cannulation and determine whether this probe enhances axillary vein imaging, accelerates the central vein cannulation procedure and reduces the rate of complications compared to the linear probe. Methods: 100 participants were recruited and allocated into two groups: the linear probe group and the hockey stick probe group. All procedures were performed by two senior anesthesia and intensive care residents, each with experience of over 100 central vascular access procedures. Follow-up chest X-rays were taken two hours post-procedure to verify the correct position of the catheter and to rule out complications such as pneumothorax, hemothorax, cardiac tamponade, and incorrect line placement.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years old
* scheduled for elective central venous catheter in the axillary vein

Exclusion Criteria:

* medical contraindication for axillary vein cannulation (coagulation abnormalities, local skin infection or chest wall deformation)
* patient consent decline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient scheduled for elective placement of the central venous catheter in the axillary vein.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Success on first attempt | 24 hours
  An attempt is defined by every needle direction change. Whenever vein puncture was not achieved by a simple, straight movement without any change of direction in any plane this cannulation was not counted as success at first attempt
Number attempts | 24 hours
  An attempt is defined by every needle direction change. Whenever vein puncture was not achieved by a simple, straight movement without any change of direction in any plane this cannulation was not counted as success at first attempt
Procedure Time | 24 hours
  The procedure time measurement stops when skin dressing is applied. Time measurement was done by an independent observer.
Cumulative number of complications | 24 hours
  Complications early and late were recorded either with ultrasonography immedi-ately after the procedure or in the chest X-ray 2 hours after.

CONTACTS AND LOCATIONS:
Locations (1):
- II Klinika Anestezjologii i Intensywnej Terapii, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No